CLINICAL TRIAL: NCT02218801
Title: A Prospective Colorectal Liver Metastasis Database With an Integrated Quality Assurance Program
Acronym: CLIMB
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: European Society of Surgical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: EORTC-1409-GITCG
Record Dates: First submitted 2014-08-07; First posted 2014-08-18 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Liver Metastasis; Colorectal Carcinoma
Keywords: Liver metastasis; Colorectal carcinoma; Unresectable; Borderline resectable; Initially unresectable
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: None Retained — whole blood, plasma, serum and left-over tissue samples from either primary tumor or liver metastasis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colorectal adenocarcinoma liver metastasis: Unresectable, borderline or initially unresectable liver metastasis from a colorectal cancer
  Interventions: Other: Evaluation of treatment for liver metastasis

INTERVENTIONS:
Other: Evaluation of treatment for liver metastasis

SUMMARY:
This prospective database has two main objectives;

* to evaluate the complication rates, 30-day and 90-day mortality from different surgical strategies for unresectable, borderline resectable or initially unresectable liver metastasis from colorectal cancer.
* to establish baseline quality parameters for different surgical strategies for unresectable, borderline and initially unresectable colorectal liver metastasis (CRLM) patients.

ELIGIBILITY:
Inclusion Criteria:

* With histologically proven colorectal adenocarcinoma with liver metastasis.
* With unresectable, borderline or initially unresectable liver metastasis from a colorectal cancer assessed by a clinician or by a multi-disciplinary tumor board (MDT).

  * Unresectable is defined as no possibility of completely resecting all tumor due to size, location or number of deposits.
  * Borderline is defined as potentially operable but technically or biologically more challenging to resect as evaluated by the MDT.
  * Initially unresectable is defined as metastasis that have been down-sized after conversion chemotherapy and evaluated by the MDT to be resectable
* discussed by a multidisciplinary team before surgery.
* Participants of the MDT must include at least one liver surgeon, one radiologist and one oncologist. They will determine the resectability of the CRLM according to local practice.
* With a possibility of a surgical procedure (resection with or without portal vein embolization, intraoperative local ablative technique or a combined approach) assessed during the MDT.
* Age ≥ 18 years.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Any psychological, familial, or sociological condition potentially hampering understanding of the research project.
* Any other malignancy other than in situ carcinoma of the cervix or non-melanoma skin cancer (unless there has been a disease-free interval of at least 5 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver metastasis of colorectal adenocarcinoma (unresectable, borderline resectable or initially unresectable)
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Number of post-operative complications | 1 year

SECONDARY OUTCOMES:
Overall survival after 2 years of follow-up | 3 years
Progression free survival at 2 years | 3 years
Number of post-operative complications in the first 50 patients compared to the second 50 patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Serge Evrard, Prof., Study Chair — Institut Bergonié; Graeme Poston, Prof., Study Chair — Aintree University Hospital
Locations (16):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Der Wiener Krankenanstaltenverbund - Krankenanstalt Rudolfstiftung, Vienna
- University Hosptial Gent, Ghent, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- France (2):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
- Germany (2):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Klinikum Der J.W. Goethe Universitaet, Frankfurt am Main
- Istituto Europeo di Oncologia, Milan, Italy
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Leiden University Medical Centre, Leiden
- Oncology Institute of Vojvodina, Kamenitz, Serbia
- Hospital De Fuenlabrada, Fuenlabrada, Spain
- Karolinska University Hospital, Stockholm, Sweden
- Hôpitaux universitaires de Genève - HUG, Geneva, Switzerland
- Aintree University Hospital NHS Trust, Liverpool, United Kingdom